CLINICAL TRIAL: NCT01516281
Title: Imaging Biomarkers of Delayed Sequelae in Mild to Moderate Traumatic Brain Injury
Brief Title: Imaging Biomarkers of Delayed Sequelae in Trauma Brain Injury
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: EH11-345
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2016-01

CONDITIONS: Traumatic Brain Injury; Parkinson's Disease
Keywords: TBI; PD
MeSH Terms: conditions — Brain Injuries, Traumatic; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collect blood and extract and store plasma and DNA from 100 mTBI and 100 mTBI- subjects undergoing clinical assessments and DaTscan studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mTBI: Historical cohort of subjects seen in the emergency rooms of NorthShore University HealthSystem with ICD-9 diagnoses of mild or moderate traumatic brain injury during the years 2006-2011 (7,122 subjects). 100 mTBI+ subjects are randomly selected for clinical assessment and DaTscan.
- mTBI-: Historical cohort of subjects seen in the emergency rooms of NorthShore University HealthSystem with ICD-9 diagnoses of disorders other than mild or moderate traumatic brain injury during the years 2006-2011 (7,122 subjects). 100 mTBI- subjects are randomly selected for clinical assessment and DaTscan.

SUMMARY:
The purpose of this study is to learn if a new brain imaging technology called DaTscan can detect subtle changes in the brain that are similar to those seen in early Parkinson's disease (PD). The results of this study may provide more information about a possible association between mild to moderate traumatic brain injury (mTBI) and PD. The objectives of this study are to define and describe a group of approximately 7,122 mTBI subjects and 7,122 subjects without mTBI (mTBI-) seen in the Emergency Rooms of NorthShore University HealthSystem during the years 2006-2011, and to select from willing eligible subjects a random sample of 100 mTBI subjects and 100 mTBI- subjects (of the same age and gender) to undergo written informed consent, neurological examinations, blood drawing for DNA extraction and storage, and DaTscan brain imaging. The investigators will compare the findings from persons who experienced mTBI (cases) to persons without a history of brain injury (mTBI- or "controls").

DETAILED DESCRIPTION:
This study is being done to learn if a new brain imaging technology called DaTscan can detect subtle changes in the brain ("biomarkers") that are similar to those seen in early Parkinson's disease (PD). The results of this study may provide more information about a potential link between mild to moderate traumatic brain injury (mTBI) and PD. We will compare findings from persons who experienced mTBI ("cases") to persons without history of brain injury (mTBI-or "controls"). This study may provide preliminary data that might be used to help design future long-term studies.

The investigators propose scientific studies with one specific aim and two hypotheses:

Specific aim: to determine if one year post emergency room (ER) visits, DaTscan uptake (Ioflupane I123 injection and single photon emission computerized tomography) is lower in subjects exposed to mTBI (defined as a closed head trauma that results in loss of consciousness or amnesia for less than 24 hours) than in subjects not exposed to mTBI (without closed head trauma; mTBI-).

Hypotheses:

Hypothesis #1: mTBI is a risk factor for Parkinson's disease (PD). Hypothesis #2: DaTscan is able to detect subclinical PD (as measured by a dopamine transporter deficiency) in mTBI subjects.

ELIGIBILITY:
Inclusion Criteria:

* mTBI or mTBI- survey respondents
* Ages 18-100 years
* Without a history of parkinsonism or tremor

Exclusion Criteria:

* History of parkinsonism or tremor
* Lugol or iodide allergy
* Contraindicated medications for DaTscan
* Pregnancy or nursing mothers
* Renal or liver impairment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A historical cohort of 7,122 mTBI cases and 7,122 age and gender matched mTBI- controls was defined from the electronic medical records of NorthShore University HealthSystem. From survey respondents we are randomly selecting 100 mTBI cases and 100 age and gender matched mTBI- controls to undergo neurological examinations and DaTscan studies.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
DaTSCAN | At least one year post ER visit for mTBI or mTBI-
  We will perform qualitative (visual) and quantitative (DaTQUANT) analyses of striatal uptake.

SECONDARY OUTCOMES:
clinical assessment | At least one year post ER visit for mTBI or mTBI-
  All subjects complete a questionnaire that documents lifelong exposures to mTBI; that screens for parkinsonism, Parkinson's disease, or tremor; and that screens for DaTSCAN exclusion criteria. We abstract medical records. Subjects eligible for DaTSCAN undergo the Montreal Cognitive Assessment (MoCA); Ohio State University TBI Identification Method Short Form (OSU-TBI-ID-SF); General Anxiety Disorder 7-item Scale (GAD7); Center for Epidemiological Studies Depression Scale (CES-D); Rivermead Post Concussion Symptoms Questionnaire; Insomnia Severity Index (ISI); World Health Organization Quality of Life-Brief Assessment (WHOQOL-BREF); Review of Systems; Past Medical History; Detailed Examination of Motor Function-Unified Parkinson's Disease Rating Scale (UPDRS part III); Neurological Examination; Syndromic Classification (parkinsonism, essential tremor, mild cognitive impairment); Differential Diagnosis of Parkinsonism (if applicable); Final Diagnosis of Parkinsonism (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Demetrius M Maraganore, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States